# **Study Protocol**

Title: "Phase II/III Clinical Trial study to evaluate efficacy and Safety of C-IVIG therapy in Severe COVID-19 Patients".

NCT04891172

Date: October 4, 2022

# **Contents**

| Title: "Phase II/III Clinical Trial study to evaluate efficacy and Safety of C-IVIG to | • • |
|---|---|
| 19 Patients" | |
| STUDY PROTOCOL | 3 |
| General Information | 3 |
| Title: "Phase II/III Clinical Trial study to evaluate efficacy and Safety of C-IVIG to 19 Patients" | • • |
| Principal and Co-Prinicipal Investigators | 3 |
| Trial Sites | 3 |
| Background Information | 3 |
| Objective | 3 |
| Trial Design | 3 |
| Participants | 4 |
| Intervention and comparator | 4 |
| Selection and Withdrawal of Subjects | 4 |
| Plasma collection from donors (recovered COVID-19 individuals): | 4 |
| Administration of C-IVIG in respective doses by medical experts in selected in | ecipient5 |
| DECODING PROCEDURES FOR BLINDED TRIALS Error! | Bookmark not defined. |

#### STUDY PROTOCOL

#### **General Information:**

Title: "Phase II/III Clinical Trial study to evaluate efficacy and Safety of C-IVIG therapy in Severe COVID-19 Patients".

## **Principal and Co-Prinicipal Investigators**

Principal Investigator: Dr. Shaukat Ali

Co- Principal Investigator: Dr. Shobha Luxmi

Co- Principal Investigator: Abdul Samad Khan

Co-Principal Investigator: Dr. Muneeba Ahsan Sayeed

#### **Trial Sites**

Dow University of Health Sciences (Ojha Campus), Karachi, Sindh

Sindh Infectious Disease Hospital and Research Center, Karachi, Sindh

PAF hospital Faisal Base, Karachi, Sindh

#### **Background Information:**

Anti-COVID19 Intravenous immunoglobulin (C-IVIg) is a mixture of IgG, IgA, IgM and Albumin derived from recovered COVID1-19 participant via Caprylic acid process. Anti-COVID19 Intravenous immunoglobulin (C-IVIg) Contain a total amount of protein 46±3.7g/L in which upto 80% is IgG, 4.0% is IgM, IgA is 15.8% and Albumin is <0.4. Anti-COVID19 C-IVIG is used in the treatment COVID 19 severe and critical patients. The dosage form is Liquid and route of administration is intravenous. The indication to given C-IVIG is PCR positive COVID 19. In non-clinical studies C-IVIG has been observed Safety and in phase I trial shown remarkable results in Safety as well as efficacy at Dow University Hospital, Karachi. 28 day mortality have been reduced markedly which were given single dose of C-IVIG intravenously with Standard of Care when compared to Control with Standard of care. It has been observe that in 28 day patient monitoring did not report any drug related serious adverse event like organ damage, disability or permanent damage.

#### **Objective**

The aim of this trial is to investigate the safety and clinical efficacy of passive immunization therapy through Hyperimmune anti-COVID-19 Intravenous Immunoglobulin (C-IVIG: 5% liquid formulation), on severe COVID-19 patients.

#### **Trial Design**

This is a phase II/III multi-centred, randomized controlled, single-blinded, superiority trial, through parallel-group design. Participants will be randomized either to receive C-IVIG and standard care or only standard care (1:1).

#### **Participants**

Consenting patients above 18 years that are classified by the treating physician as severe i.e. showing symptoms of COVID-19 pneumonia, dyspnea, respiratory rate  $\geq$ 30/min, blood oxygen saturation  $\leq$ 90%, PaO<sub>2</sub>/FiO<sub>2</sub> <300, and lung infiltrates as seen on CXR/HRCT> 50% (on  $\leq$ 15 Liters supplemental oxygen).

Critical COVID-19 patients (patients requiring mechanical ventilation) and patients given immunomodulatory drug (Tociluzumab) are excluded from study. Patients with reported IgA deficiency, autoimmune disorder, thromboembolic disorder, and allergic reaction to immunoglobulin treatment were excluded from study. Similarly, pregnant females, patients requiring two or more inotropic agents to maintain blood pressure and patients with chronic kidney injury/failure, were also excluded from the study.

## Intervention and comparator

The study consists of intervention comprising of two groups with each group containing 155 participants. All participants will receive standard hospital care which includes airway support, anti-viral medication, antibiotics, fluid resuscitation, hemodynamic support, steroids, painkillers, and anti-pyretic. Randomized test patients will receive single dose of C-IVIG in following two dosage groups:

Group 1 (Test): Severe COVID-19 patients: Single dose of 0.15g/Kg with standard hospital care

Group 2 (Comparator): Severe COVID-19 patients: only receive standard hospital care

#### **Selection and Withdrawal of Subjects**

Plasma collection from donors (recovered COVID-19 individuals):

Selection of donor according to World Health Organization (WHO) and Federal Drug Agency (FDA) guidelines

| Inclusion Criteria for Donor | Exclusion criteria for Donor |
|---|---|
| <ul> <li>a. Submitted signed consent.</li> <li>b. Eligible to donate blood.</li> <li>c. Negative for HIV, HBV, HCV, syphilis and malarial parasite.</li> <li>d. Complete resolution of symptoms at least 14</li> <li>e. days prior to donation</li> <li>f. Defined SARS-CoV-2 neutralizing antibody</li> </ul> | <ul> <li>a. Pre-existing condition Contra indicative for donating blood (HIV, viral hepatitis, tuberculosis, syphilis, oncological conditions, malaria).</li> <li>b. Bleeding tendency.</li> <li>c. Anemia.</li> <li>d. Fever of unknown origin</li> </ul> |

#### Plasma Collection

300-1000 ml plasma will be collected from consenting COVID-19 recovered patients (two weeks after resolution of symptoms) using plasmapheresis technique. Plasmapheresis is a technique where using a machine the blood components are separated, keeping the required component, in this case plasma, and returning other components like RBCs. Plasma will be stored according

to WHO guidelines. Aliquot of plasma will be screened for syphilis, malarial parasite HIV, HBV, HCV, and COVID–19 by Nucleic Acid Test (NAT). The screened stored plasma qualifying safety criteria will be pooled and fractionated to obtain Anti-COVID hyperimmune immunoglobulin.

# Administration of C-IVIG in respective doses by medical experts in selected recipient *Recipient criteria*

| Inclus | nclusion criteria for Recipient Exclusion criteria for Recipient | | sion criteria for Recipient |
|---|---|---|---|
| 1. | Above 18 years of age | a. | Critical COVID-19 patients |
| 2. | Have positive COVID PCR on | b. | Pregnant females |
| | nasopharyngeal and/or oropharyngeal | C. | Previous allergic reaction to |
| | swabs | | immunoglobulin treatment |
| 3. | classified as severe* COVID-19 according to | d. | Patient given immunomodulatory drug |
| | WHO guideline | | (e.g. tociluzumab) |
| 4. | Consent given by the patient or first | e. | Patient requiring 2 inotropic agents to |
| | degree relative | | maintain blood pressures |
| | | f. | Known case of any autoimmune disorder |
| | | g. | Chronic kidney disease |
| | | h. | Known case of thromboembolic disorder |
| | | i. | Aseptic meningitis |

<sup>\*</sup>Severe COVID-19 is defined by one or more of the following: dyspnea, respiratory frequency  $\geq$ 30/min, blood oxygen saturation  $\leq$ 90%, PaO<sub>2</sub>/FiO<sub>2</sub> ratio <300, lung infiltrates as seen through CXR/HRCT >50% (On  $\leq$ 15 Liters supplemental oxygen)